CLINICAL TRIAL: NCT00746005
Title: Challenge Study: The Efficacy of Fish Oil Supplementation on Cognitive Performance in MCI Patients and the Influence of the APOE-epsilon4 Allele
Brief Title: Efficacy of Fish Oil Supplementation on Cognition in MCI Patients and the Influence of the APOE4 Allele
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University (Other)
Collaborators: Radboud University Medical Center (Other)
Responsible Party: Lisette de Groot, Wageningen University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2008/112
Record Dates: First submitted 2008-08-30; First posted 2008-09-03 (Estimated); Last update posted 2011-01-12 (Estimated); Status verified 2011-01

CONDITIONS: Mild Cognitive Impairment
Keywords: mild cognitive impairment
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Fish Oils; Sunflower Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): 3 g EPA-DHA
  Interventions: Dietary Supplement: fish oil
- 2 (Placebo Comparator): Placebo: sunflower oil
  Interventions: Dietary Supplement: placebo, sunflower oil

INTERVENTIONS:
Dietary Supplement: fish oil — 3 g fish oil (3078 mg) total EPA 1512 mg and total DHA 1026 mg
  Arms: 1
Dietary Supplement: placebo, sunflower oil — 3 g of sunflower oil
  Arms: 2

SUMMARY:
To study the short term effects of a pharmacological dose of fish oil on cognitive performance and on cerebral blood flow. Furthermore, we want to investigate whether carriers of the APOEε4 allele respond differently to fish oil treatment compared to non-carriers.

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* Diagnosed as having amnestic MCI: based on specific memory disturbances (cut-off of 1 sd, single or multiple domain amnestic MCI, according to Busse A et al37)
* Presence of a principal caregiver willing to assist for a successful participation
* Informed consent signed

Exclusion Criteria:

* Current or recent (<4 weeks) use of fish oil supplements
* Consumption of fish more than 2 times/week
* Current use of dementia (Alzheimer) medication
* Current use of acenocoumarol or other anti-thrombotic drugs (because of the high dose of fish oil)
* Serious liver disease
* Use of more than 4 glasses of alcohol per day
* Unable to participate as judged by the responsible medical physician
* Allergy to fish(oil)
* Swallowing problems
* Participation in another clinical trial less than 2 months before the start of the trial or at the same time

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2008-10; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
cognitive performance | baseline and after 4 weeks

SECONDARY OUTCOMES:
blood flow-velocity in the middle cerebral arteries (assessed with TCD) and cortical tissue oxygenation, cerebral autoregulation, cerebral blood volume (assessed with NIRS | baseline and after 4 weeks

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - Ziekenhuis Gelderse Vallei, Ede, Gelderland
  - Radboud University Medical Center, Nijmegen, Gelderland

REFERENCES:
- See also: Related Info — http://www.humannutrition.nl